CLINICAL TRIAL: NCT03342898
Title: A Randomized, Observer-Blind, Placebo-Controlled, Phase 3 Trial to Investigate the Immunogenicity and Safety of a Tetravalent Dengue Vaccine Candidate and a Yellow Fever YF-17D Vaccine Administered Concomitantly and Sequentially in Healthy Subjects Aged 18 to 60 Years in Non-Endemic Country(Ies)
Brief Title: Immunogenicity and Safety of Tetravalent Dengue Vaccine (TDV) Administered With a Yellow Fever Vaccine in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DEN-305; U1111-1201-5257 (Registry Identifier: WHO)
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Dengue
Keywords: Drug Therapy
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: YF-17D + Placebo/TDV/TDV (Experimental): YF-17D vaccine, 0.5 mL injection, subcutaneously (SC) plus YF 17D + TDV placebo-matching 0.5 mL, injection, SC on Day 1, followed by TDV, 0.5 mL, injection, SC on Day 90 (first dose), followed by TDV, 0.5 mL, injection, SC on Day 180 (second dose).
  Interventions: Biological: YF-17D; Biological: TDV; Drug: Placebo
- Group 2: TDV + Placebo/TDV/YF-17D (Experimental): TDV, 0.5 mL, injection, SC plus TDV placebo-matching, 0.5 mL injection, SC on Day 1 (first dose), followed by TDV, 0.5 mL, injection, SC on Day 90 (second dose), followed by YF-17D vaccine, 0.5 mL, injection, SC on Day 180.
  Interventions: Biological: YF-17D; Biological: TDV; Drug: Placebo
- Group 3: TDV + YF-17D/TDV/Placebo (Experimental): TDV, 0.5 mL, injection, SC plus YF-17D vaccine, 0.5 mL, injection, SC on Day 1 (first dose), followed by TDV, 0.5 mL, injection, SC on day 90 (second dose), followed by TDV + YF 17D placebo-matching, 0.5 mL, injection, SC on Day 180.
  Interventions: Biological: YF-17D; Biological: TDV; Drug: Placebo

INTERVENTIONS:
Biological: YF-17D — YF-17D SC injection.
Biological: TDV — TDV SC injection.
  Other Names: TAK-003; DENVax
Drug: Placebo — Normal Saline (0.9% NaCl) SC injection.

SUMMARY:
The main purpose of this study is to assess the immunogenicity and safety of the concomitant and sequential administration of yellow fever (YF) vaccine and tetravalent dengue vaccine (TDV) in healthy participants aged 18 to 60 years living in country non-endemic for both dengue and YF.

DETAILED DESCRIPTION:
The vaccine tested in this study is TDV also known as TAK-003 (DENVax). TDV with concomitant and sequential administration of yellow fever (YF-17D) vaccine will be tested to assess immunogenicity and safety in healthy adult participants in non-endemic area(s) for both dengue and YF.

The study will enroll 900 healthy participants. Participants will be randomized to 3 groups in 1:1:1 ratio and will be administered concomitantly and sequentially. The 3 groups are:

* Group 1: YF-17D vaccine + placebo concomitantly administered on Day 1, first dose of TDV administered on Day 90 and second dose of TDV administered on Day 180.
* Group 2: first dose of TDV + placebo concomitantly administered on Day 1, second dose of TDV administered on Day 90 and YF-17D vaccine administered on Day 180.
* Group 3: first dose of TDV + YF-17D vaccine concomitantly administered on Day 1, second dose of TDV administered on Day 90 and placebo administered on Day 180.

This multi-center trial will be conducted in the United States. The overall time to participate in this study is 360 days. Participants will make multiple visits to the clinic with a 6-month follow up including a final visit at Day 360 for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Is aged 18 to 60 years inclusive, at the time of randomization.
2. Is in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs), and the clinical judgment of the Investigator.

Exclusion Criteria:

1. Has an elevated oral temperature ≥ 38°C (100.4°F) within 3 days of the intended date of vaccination.
2. Has contraindications, warnings and/or precautions to vaccination with the YF-17D vaccine as specified within the product information (especially history of thymus dysfunction).
3. Female participant who are pregnant or breastfeeding
4. Has any history of progressive or severe neurologic disorder, seizure disorder or neuro-inflammatory disease (e.g., Guillain-Barre syndrome) or suspected impairment/alteration of immune function.
5. Has body mass index (BMI) greater than or equal to 35 kg/m^2 (=weight in kg/[height in meters^2]).
6. Is intent to travel to dengue or YF endemic countries during the trial period.
7. Has received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this trial or who are planning to receive any non-trial vaccine within 28 days of trial vaccine administration.
8. Has previous and planned vaccination (during the trial conduct), against any flavivirus including dengue, YF, Japanese encephalitis (JE) or tick-borne encephalitis viruses.
9. Has previous participation in any clinical trial of a dengue or other flavivirus (e.g., West Nile [WN] virus) candidate vaccine, except for participants who received placebo in those trials.
10. Has a current or previous infection with a flavivirus such as dengue, Zika, YF, JE, WN fever, or Saint Louis encephalitis viruses and participants with a history of prolonged (≥1 year) habitation in a dengue endemic area.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 900 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2019-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (11):
- United States (11):
  - Coastal Clinical Research Inc, Mobile, Alabama
  - Empire Clinical Research, Pomona, California
  - Advanced Clinical Research, Meridian, Idaho
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - Meridian Clinical Research LLC, Omaha, Nebraska
  - Regional Clinical Research Inc., Endwell, New York
  - Rapid Medical Research Inc, Cleveland, Ohio
  - Tekton Research, Austin, Texas
  - Advanced Clinical Research, West Jordan, Utah
  - Clinical Research Associates of Tidewater, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Rauscher M, Youard Z, Faccin A, Patel SS, Pang H, Zent O. Pregnancy outcomes following unintentional exposure to TAK-003, a live-attenuated tetravalent dengue vaccine. Expert Rev Vaccines. 2025 Dec;24(1):221-229. doi: 10.1080/14760584.2025.2480297. Epub 2025 Mar 27. PMID 40099800
- [Derived] Tricou V, Essink B, Ervin JE, Turner M, Escudero I, Rauscher M, Brose M, Lefevre I, Borkowski A, Wallace D. Immunogenicity and safety of concomitant and sequential administration of yellow fever YF-17D vaccine and tetravalent dengue vaccine candidate TAK-003: A phase 3 randomized, controlled study. PLoS Negl Trop Dis. 2023 Mar 8;17(3):e0011124. doi: 10.1371/journal.pntd.0011124. eCollection 2023 Mar. PMID 36888687

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 11 investigative sites in the United States from 28 Feb 2018 to 22 May 2019.
Pre-assignment Details: Healthy participants were enrolled in 1:1:1 ratio in 3 parallel groups. Participants received concomitant and sequential administration of yellow fever (YF) vaccine and tetravalent dengue vaccine (TDV) in Groups 1, 2 and 3.
Period: Overall Study
Arm/Group | Group 1: YF-17D + Placebo/TDV/TDV | Group 2: TDV + Placebo/TDV/YF-17D | Group 3: TDV + YF-17D/TDV/Placebo
Started | 300 | 300 | 300
Completed | 246 | 247 | 246
Not Completed | 54 | 53 | 54
Not completed — Adverse Event | 3 | 1 | 0
Not completed — Lost to Follow-up | 44 | 40 | 42
Not completed — Withdrawal of Consent | 5 | 9 | 11
Not completed — Death | 0 | 1 | 1
Not completed — Reason not Specified | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set included all randomized participants who received at least 1 dose of the trial vaccines.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: YF-17D + Placebo/TDV/TDV | Group 2: TDV + Placebo/TDV/YF-17D | Group 3: TDV + YF-17D/TDV/Placebo | Total
Number analyzed (Participants) | 300 | 300 | 300 | 900
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (12.41) | 40.0 (12.91) | 41.4 (12.67) | 41.0 (12.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167 | 170 | 176 | 513
  Male | 133 | 130 | 124 | 387
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 25 | 31 | 82
  Not Hispanic or Latino | 272 | 270 | 266 | 808
  Unknown or Not Reported | 2 | 5 | 3 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 2 | 7
  Asian | 3 | 4 | 7 | 14
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 1 | 3
  Black or African American | 77 | 103 | 84 | 264
  White | 205 | 186 | 201 | 592
  More than one race | 5 | 0 | 2 | 7
  Unknown or Not Reported | 5 | 5 | 3 | 13
Height [Mean (Standard Deviation); unit: cm] | 171.3 (9.29) | 170.1 (9.05) | 170.5 (8.85) | 170.6 (9.07)
Weight [Mean (Standard Deviation); unit: kg] | 82.40 (15.40) | 78.52 (14.65) | 80.87 (16.94) | 80.60 (15.75)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI = Weight(kg)/height(m)^2.
  kg/m^2 | 28.00 (4.29) | 27.07 (4.30) | 27.66 (4.49) | 27.58 (4.37)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Are YF and Dengue Virus (DENV)-Naive at Baseline and Are Seroprotected Against YF on Day 30 as Measured by Plaque Reduction Neutralization Test (PRNT)
Description: Seroprotection was defined as reciprocal anti-YF neutralizing antibody titer ≥10. Immunological naivety to YF and DENV was defined as Baseline reciprocal neutralizing antibody titers <10 for YF and for the 4 dengue serotypes. The 95% CI was calculated using exact Clopper-Pearson method.
Time Frame: Day 30
Population: Yellow Fever Per-Protocol Set (YF PPS) included all participants YF and DENV-naïve at Baseline who received >=1 dose of trial vaccine, with data available for Baseline and Day 30, and who had no major protocol violations. Overall number analyzed are participants with data available for analyses at given time point within pre-specified visit window.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: YF-17D + Placebo/TDV/TDV | Group 2: TDV + Placebo/TDV/YF-17D | Group 3: TDV + YF-17D/TDV/Placebo
Number analyzed (Participants) | 211 | 234 | 229
percentage of participants | 99.5 [97.4 to 100.0] | 9.8 [6.3 to 14.4] | 99.1 [96.9 to 99.9]
Statistical Analysis 1: Comparison: Group 1: YF-17D + Placebo/TDV/TDV vs Group 3: TDV + YF-17D/TDV/Placebo; Test type: Non-Inferiority — Non-inferiority of the immune response was performed only between YF + TDV (Group 3) and YF + Placebo (Group 1) at Day 120. Non-inferiority between Group 3 and Group 1 was concluded if the upper bound of the 95% CI for the seroprotection rate difference (Group 1 - Group 3) was less than 5%; Seroprotection Rate Difference = 0.40, 95% CI 2-sided [-1.85 to 2.69] — The Newcombe score method was used to compute the 95% CI of the seroprotection rate difference

2. Secondary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibodies for Each of the 4 Dengue Serotypes on Days 30, 90, 120, 180 and 210 in Participants YF and DENV-naive at Baseline
Description: GMTs of neutralizing antibodies was measured by microneutralization test 50% [MNT50] for each of the 4 dengue serotypes. The 4 DENV serotypes are DENV-1, DENV-2, DENV-3 and DENV-4.
Time Frame: Pre-second and -third vaccination (Days 90 and 180, respectively); and 1 month post -first, second, and third vaccination (Days 30, 120, and 210, respectively)
Population: Per-Protocol Set (PPS) included all participants YF and DENV-naïve at Baseline who received >=1 dose of trial vaccine, with data available for Baseline and >=1 post-Baseline immunogenicity measurement, and who had no major protocol violations.Number analyzed are participants with data available at given time point within pre-specified visit window.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: YF-17D + Placebo/TDV/TDV | Group 2: TDV + Placebo/TDV/YF-17D | Group 3: TDV + YF-17D/TDV/Placebo
Number analyzed (Participants) | 192 | 208 | 189
titer
  Day 30, DENV-1: number analyzed (Participants) | 184 | 193 | 185
  Day 30, DENV-1 | 6.0 [5.4 to 6.7] | 226.2 [178.7 to 286.4] | 119.4 [93.0 to 153.4]
  Day 30, DENV-2: number analyzed (Participants) | 184 | 193 | 185
  Day 30, DENV-2 | 7.7 [6.6 to 9.0] | 5431.1 [3930.2 to 7505.3] | 650.8 [438.1 to 966.7]
  Day 30, DENV-3: number analyzed (Participants) | 184 | 193 | 185
  Day 30, DENV-3 | 5.8 [5.2 to 6.4] | 172.0 [129.4 to 228.5] | 70.9 [54.1 to 92.9]
  Day 30, DENV-4: number analyzed (Participants) | 184 | 193 | 185
  Day 30, DENV-4 | 6.1 [5.4 to 6.9] | 142.0 [108.7 to 185.4] | 49.8 [39.3 to 63.1]
  Day 90, DENV-1 | 6.0 [5.5 to 6.6] | 147.5 [114.6 to 189.7] | 95.1 [74.0 to 122.2]
  Day 90, DENV-2 | 7.8 [6.6 to 9.2] | 2846.5 [2273.6 to 3563.7] | 1547.2 [1198.1 to 1998.0]
  Day 90, DENV-3 | 5.9 [5.3 to 6.5] | 73.1 [58.3 to 91.7] | 70.1 [57.3 to 85.7]
  Day 90, DENV-4 | 5.9 [5.3 to 6.4] | 56.1 [45.0 to 70.0] | 49.1 [41.0 to 58.8]
  Day 120, DENV-1: number analyzed (Participants) | 175 | 198 | 177
  Day 120, DENV-1 | 403.9 [335.3 to 486.6] | 297.1 [239.8 to 368.1] | 182.6 [145.5 to 229.2]
  Day 120, DENV-2: number analyzed (Participants) | 175 | 198 | 177
  Day 120, DENV-2 | 4691.3 [3688.6 to 5966.4] | 2616.1 [2133.1 to 3208.4] | 1947.7 [1639.9 to 2313.2]
  Day 120, DENV-3: number analyzed (Participants) | 175 | 198 | 177
  Day 120, DENV-3 | 636.4 [525.6 to 770.5] | 131.4 [110.5 to 156.3] | 104.5 [87.9 to 124.1]
  Day 120, DENV-4: number analyzed (Participants) | 175 | 198 | 177
  Day 120, DENV-4 | 678.5 [568.7 to 809.4] | 111.8 [94.5 to 132.1] | 97.7 [81.4 to 117.3]
  Day 180, DENV-1 | 251.4 [209.0 to 302.3] | 227.0 [177.4 to 290.4] | 147.0 [115.8 to 186.6]
  Day 180, DENV-2 | 2413.5 [2038.6 to 2857.3] | 1959.3 [1584.1 to 2423.5] | 1800.0 [1535.8 to 2109.7]
  Day 180, DENV-3 | 342.3 [294.6 to 397.9] | 84.9 [70.1 to 102.8] | 75.8 [65.2 to 88.3]
  Day 180, DENV-4 | 358.4 [302.8 to 424.2] | 83.7 [69.9 to 100.3] | 69.6 [59.0 to 82.3]
  Day 210, DENV-1: number analyzed (Participants) | 171 | 187 | 176
  Day 210, DENV-1 | 267.5 [221.5 to 323.2] | 679.9 [549.7 to 841.0] | 138.2 [108.3 to 176.2]
  Day 210, DENV-2: number analyzed (Participants) | 171 | 187 | 176
  Day 210, DENV-2 | 2248.0 [1902.3 to 2656.6] | 3798.1 [3139.4 to 4595.0] | 1688.0 [1431.7 to 1990.1]
  Day 210, DENV-3: number analyzed (Participants) | 171 | 187 | 176
  Day 210, DENV-3 | 301.8 [262.7 to 346.6] | 406.4 [345.4 to 478.1] | 64.3 [54.3 to 76.2]
  Day 210, DENV-4: number analyzed (Participants) | 171 | 187 | 176
  Day 210, DENV-4 | 347.4 [297.5 to 405.6] | 436.5 [374.7 to 508.5] | 56.6 [46.9 to 68.2]
Statistical Analysis 1: Comparison: Group 2: TDV + Placebo/TDV/YF-17D vs Group 3: TDV + YF-17D/TDV/Placebo; Day 120, DENV-1; Test type: Non-Inferiority — Non-inferiority of the immune response was performed only between TDV + YF (Group 3) and TDV + Placebo (Group 2) at Day 120. Non-inferiority between Group 3 and Group 2 was concluded if the upper bound of the 95% CI for the GMT ratio (Group 2/Group 3) was less than 2.0; Geometric Mean Ratio = 1.6, 95% CI 2-sided [1.19 to 2.22] — Analysis of variance (ANOVA) model was used for analysis, including log-transformed value of titer as the dependent variable and trial group as a factor
Statistical Analysis 2: Comparison: Group 2: TDV + Placebo/TDV/YF-17D vs Group 3: TDV + YF-17D/TDV/Placebo; Day 120, DENV-2; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio = 1.3, 95% CI [1.03 to 1.75] — ANOVA model was used for analysis, including log-transformed value of titer as the dependent variable and trial group as a factor
Statistical Analysis 3: Comparison: Group 2: TDV + Placebo/TDV/YF-17D vs Group 3: TDV + YF-17D/TDV/Placebo; Day 120, DENV-3; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio = 1.3, 95% CI [0.99 to 1.61] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 4: Comparison: Group 2: TDV + Placebo/TDV/YF-17D vs Group 3: TDV + YF-17D/TDV/Placebo; Day 120, DENV-4; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio = 1.1, 95% CI 2-sided [0.89 to 1.46] — [estimate comment as in outcome 2, analysis 2]

3. Secondary Outcome: Percentage of Participants Who Are Seropositive for Each of the 4 Dengue Serotypes on Days 30, 90, 120, 180 and 210 in Participants YF and DENV-naive at Baseline
Description: Seropositivity rate was defined as the percentage of seropositive participants as derived from the titers of dengue-neutralizing antibodies. Seropositivity was defined as a reciprocal neutralizing titer ≥10. Seropositivity for each dengue serotype were analyzed and was summarized as: DENV-1, DENV-2, DENV-3, and DENV-4.
Time Frame: Pre-second and -third vaccination (Days 90 and 180, respectively); and 1-month post -first, -second, and -third vaccination (Days 30, 120, and 210, respectively)
Population: PPS included all participants YF and DENV-naïve at Baseline who received >=1 dose of trial vaccine, with data available for Baseline and >=1 post-Baseline immunogenicity measurement, and who had no major protocol violations. Number analyzed are participants with data available at given time point within pre-specified visit window.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: YF-17D + Placebo/TDV/TDV | Group 2: TDV + Placebo/TDV/YF-17D | Group 3: TDV + YF-17D/TDV/Placebo
Number analyzed (Participants) | 192 | 208 | 189
percentage of participants
  Day 30, DENV-1: number analyzed (Participants) | 184 | 193 | 185
  Day 30, DENV-1 | 6.5 [3.4 to 11.1] | 93.3 [88.8 to 96.4] | 87.6 [81.9 to 92.0]
  Day 30, DENV-2: number analyzed (Participants) | 184 | 193 | 185
  Day 30, DENV-2 | 15.8 [10.8 to 21.8] | 95.9 [92.0 to 98.2] | 88.1 [82.6 to 92.4]
  Day 30, DENV-3: number analyzed (Participants) | 184 | 193 | 185
  Day 30, DENV-3 | 4.3 [1.9 to 8.4] | 88.1 [82.7 to 92.3] | 80.5 [74.1 to 86.0]
  Day 30, DENV-4: number analyzed (Participants) | 184 | 193 | 185
  Day 30, DENV-4 | 7.1 [3.8 to 11.8] | 89.6 [84.4 to 93.6] | 78.4 [71.7 to 84.1]
  Day 90, DENV-1 | 8.3 [4.8 to 13.2] | 90.4 [85.5 to 94.0] | 89.4 [84.1 to 93.4]
  Day 90, DENV-2 | 14.6 [9.9 to 20.4] | 97.1 [93.8 to 98.9] | 94.2 [89.8 to 97.1]
  Day 90, DENV-3 | 5.7 [2.9 to 10.0] | 84.6 [79.0 to 89.2] | 90.5 [85.4 to 94.3]
  Day 90, DENV-4 | 6.3 [3.3 to 10.7] | 84.6 [79.0 to 89.2] | 89.4 [84.1 to 93.4]
  Day 120, DENV-1: number analyzed (Participants) | 175 | 198 | 177
  Day 120, DENV-1 | 99.4 [96.9 to 100.0] | 99.5 [97.2 to 100.0] | 99.4 [96.9 to 100.0]
  Day 120, DENV-2: number analyzed (Participants) | 175 | 198 | 177
  Day 120, DENV-2 | 99.4 [96.9 to 100.0] | 98.5 [95.6 to 99.7] | 99.4 [96.9 to 100.0]
  Day 120, DENV-3: number analyzed (Participants) | 175 | 198 | 177
  Day 120, DENV-3 | 98.9 [95.9 to 99.9] | 98.5 [95.6 to 99.7] | 98.3 [95.1 to 99.6]
  Day 120, DENV-4: number analyzed (Participants) | 175 | 198 | 177
  Day 120, DENV-4 | 99.4 [96.9 to 100.0] | 99.0 [96.4 to 99.9] | 97.7 [94.3 to 99.4]
  Day 180, DENV-1 | 99.0 [96.3 to 99.9] | 97.1 [93.8 to 98.9] | 95.8 [91.8 to 98.2]
  Day 180, DENV-2 | 100.0 [98.1 to 100.0] | 97.6 [94.5 to 99.2] | 99.5 [97.1 to 100.0]
  Day 180, DENV-3 | 99.5 [97.1 to 100.0] | 92.8 [88.4 to 95.9] | 96.3 [92.5 to 98.5]
  Day 180, DENV-4 | 99.0 [96.3 to 99.9] | 96.6 [93.2 to 98.6] | 96.8 [93.2 to 98.8]
  Day 210, DENV-1: number analyzed (Participants) | 171 | 187 | 176
  Day 210, DENV-1 | 100.0 [97.9 to 100.0] | 99.5 [97.1 to 100.0] | 96.6 [92.7 to 98.7]
  Day 210, DENV-2: number analyzed (Participants) | 171 | 187 | 176
  Day 210, DENV-2 | 100.0 [97.9 to 100.0] | 99.5 [97.1 to 100.0] | 99.4 [96.9 to 100.0]
  Day 210, DENV-3: number analyzed (Participants) | 171 | 187 | 176
  Day 210, DENV-3 | 100.0 [97.9 to 100.0] | 99.5 [97.1 to 100.0] | 93.2 [88.4 to 96.4]
  Day 210, DENV-4: number analyzed (Participants) | 171 | 187 | 176
  Day 210, DENV-4 | 99.4 [96.8 to 100.0] | 99.5 [97.1 to 100.0] | 94.3 [89.8 to 97.2]

4. Secondary Outcome: Percentage of Participants Who Are Seropositive for Multiple (2, 3 or 4) Dengue Serotypes on Days 30, 90, 120, 180 and 210 in Participants YF and DENV-naive at Baseline
Description: Seropositivity rate was defined as the percentage of seropositive participants, as derived from the titers of dengue-neutralizing antibodies. Seropositivity was defined as a reciprocal neutralizing titer ≥10. Seropositivity for multiple dengue serotypes were summarized in the following categories: at least bivalent, at least trivalent and tetravalent.
Time Frame: Pre-second and -third vaccination (Days 90 and 180, respectively); and 1-month post -first, second, and -third vaccination (Days 30, 120, and 210, respectively)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: YF-17D + Placebo/TDV/TDV | Group 2: TDV + Placebo/TDV/YF-17D | Group 3: TDV + YF-17D/TDV/Placebo
Number analyzed (Participants) | 192 | 208 | 189
percentage of participants
  Day 30, At Least Bivalent: number analyzed (Participants) | 184 | 193 | 185
  Day 30, At Least Bivalent | 5.4 [2.6 to 9.8] | 96.9 [93.4 to 98.9] | 90.8 [85.7 to 94.6]
  Day 30, At Least Trivalent: number analyzed (Participants) | 184 | 193 | 185
  Day 30, At Least Trivalent | 4.9 [2.3 to 9.1] | 91.7 [86.9 to 95.2] | 81.6 [75.3 to 86.9]
  Day 30, Tetravalent: number analyzed (Participants) | 184 | 193 | 185
  Day 30, Tetravalent | 3.8 [1.5 to 7.7] | 79.3 [72.9 to 84.8] | 65.9 [58.6 to 72.7]
  Day 90, At Least Bivalent | 6.3 [3.3 to 10.7] | 95.7 [91.9 to 98.0] | 94.7 [90.5 to 97.4]
  Day 90, At Least Trivalent | 5.7 [2.9 to 10.0] | 87.0 [81.7 to 91.3] | 88.9 [83.5 to 93.0]
  Day 90, Tetravalent | 5.7 [2.9 to 10.0] | 75.5 [69.1 to 81.2] | 82.0 [75.8 to 87.2]
  Day 120, At Least Bivalent: number analyzed (Participants) | 175 | 198 | 177
  Day 120, At Least Bivalent | 99.4 [96.9 to 100.0] | 99.5 [97.2 to 100.0] | 99.4 [96.9 to 100.0]
  Day 120, At Least Trivalent: number analyzed (Participants) | 175 | 198 | 177
  Day 120, At Least Trivalent | 99.4 [96.9 to 100.0] | 99.5 [97.2 to 100.0] | 98.3 [95.1 to 99.6]
  Day 120, Tetravalent: number analyzed (Participants) | 175 | 198 | 177
  Day 120, Tetravalent | 98.9 [95.9 to 99.9] | 97.0 [93.5 to 98.9] | 97.7 [94.3 to 99.4]
  Day 180, At Least Bivalent | 99.5 [97.1 to 100.0] | 99.0 [96.6 to 99.9] | 98.9 [96.2 to 99.9]
  Day 180, At Least Trivalent | 99.0 [96.3 to 99.9] | 97.6 [94.5 to 99.2] | 98.4 [95.4 to 99.7]
  Day 180, Tetravalent | 99.0 [96.3 to 99.9] | 88.0 [82.8 to 92.1] | 91.5 [86.6 to 95.1]
  Day 210, At Least Bivalent: number analyzed (Participants) | 171 | 187 | 176
  Day 210, At Least Bivalent | 100.0 [97.9 to 100.0] | 99.5 [97.1 to 100.0] | 98.9 [96.0 to 99.9]
  Day 210, At Least Trivalent: number analyzed (Participants) | 171 | 187 | 176
  Day 210, At Least Trivalent | 100.0 [97.9 to 100.0] | 99.5 [97.1 to 100.0] | 96.0 [92.0 to 98.4]
  Day 210, Tetravalent: number analyzed (Participants) | 171 | 187 | 176
  Day 210, Tetravalent | 99.4 [96.8 to 100.0] | 99.5 [97.1 to 100.0] | 89.2 [83.7 to 93.4]

5. Secondary Outcome: Percentage of YF and DENV-naive Participants at Baseline Who Are Seroprotected Against YF on Day 210 as Measured by PRNT
Description: Seroprotection was defined as reciprocal anti-YF neutralizing antibody titer ≥10.
Time Frame: 1-month post third vaccination (Day 210)
Population: PPS included all participants YF and DENV-naïve at Baseline who received >=1 dose of trial vaccine, with data available for Baseline and >=1 post-Baseline immunogenicity measurement, and who had no major protocol violations. Overall number analyzed: participants with data available for analyses at given time point within pre-specified visit window.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: YF-17D + Placebo/TDV/TDV | Group 2: TDV + Placebo/TDV/YF-17D | Group 3: TDV + YF-17D/TDV/Placebo
Number analyzed (Participants) | 171 | 188 | 176
percentage of participants | 100.0 [97.9 to 100.0] | 98.4 [95.4 to 99.7] | 98.9 [96.0 to 99.9]

6. Secondary Outcome: Geometric Mean Titers (GMTs) of Anti-YF Neutralizing Antibodies at Day 30 in Participants YF and DENV-Naive at Baseline
Description: Geometric mean titers of YF neutralizing antibodies was measured by plaque reduction neutralization test.
Time Frame: 1-month post-first vaccination (Day 30)
Population: YF PPS included all participants YF and DENV-naïve at Baseline who received >=1 dose of trial vaccine, with data available for Baseline and Day 30, and who had no major protocol violations. Overall number analyzed are participants with data available for analyses at given time point within pre-specified visit window.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: YF-17D + Placebo/TDV/TDV | Group 2: TDV + Placebo/TDV/YF-17D | Group 3: TDV + YF-17D/TDV/Placebo
Number analyzed (Participants) | 211 | 234 | 229
titer | 4245.7 [3526.5 to 5111.6] | 6.0 [5.5 to 6.6] | 4321.7 [3652.5 to 5113.6]
Statistical Analysis 1: Comparison: Group 1: YF-17D + Placebo/TDV/TDV vs Group 3: TDV + YF-17D/TDV/Placebo; Test type: Non-Inferiority — Non-inferiority of the immune response was performed only between YF + TDV (Group 3) and YF + Placebo (Group 1) at Day 30. Non-inferiority between Group 3 and Group 1 was concluded if the upper bound of the 95% CI for the GMT ratio (Group 1/Group 3) was less than 2.0; Geometric Mean Ratio = 1.0, 95% CI 2-sided [0.77 to 1.26] — ANOVA model was used for analyses, including the log-transformed value of titer as the dependent variable and trial group as a factor

7. Secondary Outcome: Geometric Mean Titers (GMTs) of Anti-YF Neutralizing Antibodies at Day 210 in Participants YF and DENV-Naive at Baseline
Description: Geometric mean titers of YF neutralizing antibodies was measured by plaque reduction neutralization test.
Time Frame: 1-month post-third vaccination (Day 210)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: YF-17D + Placebo/TDV/TDV | Group 2: TDV + Placebo/TDV/YF-17D | Group 3: TDV + YF-17D/TDV/Placebo
Number analyzed (Participants) | 171 | 188 | 176
titer | 2341.6 [1938.2 to 2829.0] | 3078.2 [2452.0 to 3864.4] | 1089.1 [888.1 to 1335.7]

8. Secondary Outcome: Percentage of Participants With Solicited Local (Injection Site) Adverse Events (AEs) Following Each Vaccination Dose by Severity
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a trial vaccine; it does not necessarily have to have a causal relationship with trial vaccine administration. Solicited local injection site AEs recorded from participant's-diary. Severity grade at injection site for pain: Grade 0 (No Pain), 1 (did not interfere with daily activity), 2 (interference with daily activity with or without treatment) and 3 (prevents daily activity with or without treatment). For erythema: grade 0 (<25 mm), 1 (>25-≤50 mm), 2 (>50-≤100 mm) and 3 (>100 mm). For swelling: grade 0 (<25 mm), 1 (>25-≤50 mm), 2 (>50-≤100 mm) and 3 (>100 mm). Percentages were rounded off for each category. For the first vaccination (Vac.) YF is given in Arm 1 (A1) and TDV is given in Arm 2 (A2). A1 = YF for Group 1, Placebo for Group 2, and YF for Group 3; A2 = Placebo for Group 1, TDV for Group 2, and TDV for Group 3.
Time Frame: Within 7 Days of each Vaccination (day of vaccination + 6 days)
Population: Safety Set included all randomized participants who received at least 1 dose of the trial vaccines. Number analyzed are participants with data available for the category. Only categories with at least one participant are reported.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: YF-17D + Placebo/TDV/TDV | Group 2: TDV + Placebo/TDV/YF-17D | Group 3: TDV + YF-17D/TDV/Placebo
Number analyzed (Participants) | 300 | 300 | 300
percentage of participants
  After Vac. 1, Any Local AEs, A1: number analyzed (Participants) | 289 | 285 | 282
  After Vac. 1, Any Local AEs, A1 | 13.1 | 16.8 | 27.3
  After Vac. 1, Any Local AEs, A2: number analyzed (Participants) | 289 | 285 | 282
  After Vac. 1, Any Local AEs, A2 | 13.1 | 44.2 | 48.9
  After Vac. 1, Pain: Any Severity, A1: number analyzed (Participants) | 289 | 285 | 282
  After Vac. 1, Pain: Any Severity, A1 | 12.1 | 16.5 | 24.1
  After Vac. 1, Pain: Any Severity, A2: number analyzed (Participants) | 289 | 285 | 282
  After Vac. 1, Pain: Any Severity, A2 | 12.8 | 40.0 | 42.2
  After Vac. 1, Pain: Mild, A1: number analyzed (Participants) | 289 | 285 | 282
  After Vac. 1, Pain: Mild, A1 | 9.0 | 13.7 | 21.3
  After Vac. 1, Pain: Mild, A2: number analyzed (Participants) | 289 | 285 | 282
  After Vac. 1, Pain: Mild, A2 | 10.0 | 35.1 | 34.0
  After Vac. 1, Pain: Moderate, A1: number analyzed (Participants) | 289 | 285 | 282
  After Vac. 1, Pain: Moderate, A1 | 3.1 | 2.5 | 2.1
  After Vac. 1, Pain: Moderate, A2: number analyzed (Participants) | 289 | 285 | 282
  After Vac. 1, Pain: Moderate, A2 | 2.4 | 4.6 | 6.7
  After Vac. 1, Pain: Severe, A1: number analyzed (Participants) | 289 | 285 | 282
  After Vac. 1, Pain: Severe, A1 | 0 | 0.4 | 0.7
  After Vac. 1, Pain: Severe, A2: number analyzed (Participants) | 289 | 285 | 282
  After Vac. 1, Pain: Severe, A2 | 0.3 | 0.4 | 1.4
  After Vac. 1, Erythema: Any Severity, A1: number analyzed (Participants) | 288 | 284 | 282
  After Vac. 1, Erythema: Any Severity, A1 | 2.4 | 1.8 | 3.9
  After Vac. 1, Erythema: Any Severity, A2: number analyzed (Participants) | 288 | 285 | 282
  After Vac. 1, Erythema: Any Severity, A2 | 0.7 | 19.6 | 19.5
  After Vac. 1,Erythema:Mild:2.5-5(cm), A1: number analyzed (Participants) | 288 | 284 | 282
  After Vac. 1,Erythema:Mild:2.5-5(cm), A1 | 1.7 | 1.8 | 3.9
  After Vac. 1,Erythema:Mild:2.5-5(cm), A2: number analyzed (Participants) | 288 | 285 | 282
  After Vac. 1,Erythema:Mild:2.5-5(cm), A2 | 0 | 17.5 | 18.8
  After Vac. 1,Erythema:Moderate:>5-<=10(cm), A1: number analyzed (Participants) | 288 | 284 | 282
  After Vac. 1,Erythema:Moderate:>5-<=10(cm), A1 | 0.3 | 0 | 0
  After Vac. 1,Erythema:Moderate:>5-<=10(cm), A2: number analyzed (Participants) | 288 | 285 | 282
  After Vac. 1,Erythema:Moderate:>5-<=10(cm), A2 | 0.7 | 1.8 | 0.4
  After Vac. 1,Erythema:Severe:>10(cm), A1: number analyzed (Participants) | 288 | 284 | 282
  After Vac. 1,Erythema:Severe:>10(cm), A1 | 0.3 | 0 | 0
  After Vac. 1,Erythema:Severe:>10(cm), A2: number analyzed (Participants) | 288 | 285 | 282
  After Vac. 1,Erythema:Severe:>10(cm), A2 | 0 | 0 | 0.4
  After Vac. 1, Erythema: Missing Severity, A2: number analyzed (Participants) | 288 | 285 | 282
  After Vac. 1, Erythema: Missing Severity, A2 | 0 | 0.4 | 0
  After Vac. 1, Swelling: Any Severity, A1: number analyzed (Participants) | 287 | 285 | 282
  After Vac. 1, Swelling: Any Severity, A1 | 0.7 | 1.1 | 2.1
  After Vac. 1, Swelling: Any Severity, A2: number analyzed (Participants) | 287 | 285 | 282
  After Vac. 1, Swelling: Any Severity, A2 | 0.3 | 4.2 | 5.3
  After Vac. 1,Swelling:Mild:2.5-5(cm), A1: number analyzed (Participants) | 287 | 285 | 282
  After Vac. 1,Swelling:Mild:2.5-5(cm), A1 | 0.3 | 1.1 | 1.8
  After Vac. 1,Swelling:Mild:2.5-5(cm), A2: number analyzed (Participants) | 287 | 285 | 282
  After Vac. 1,Swelling:Mild:2.5-5(cm), A2 | 0 | 4.2 | 4.6
  After Vac. 1,Swelling:Moderate:>5-<=10(cm), A1: number analyzed (Participants) | 287 | 285 | 282
  After Vac. 1,Swelling:Moderate:>5-<=10(cm), A1 | 0 | 0 | 0.4
  After Vac. 1,Swelling:Moderate:>5-<=10(cm), A2: number analyzed (Participants) | 287 | 285 | 282
  After Vac. 1,Swelling:Moderate:>5-<=10(cm), A2 | 0.3 | 0 | 0.4
  After Vac. 1,Swelling:Severe:>10(cm), A1: number analyzed (Participants) | 287 | 285 | 282
  After Vac. 1,Swelling:Severe:>10(cm), A1 | 0.3 | 0 | 0
  After Vac. 1,Swelling:Severe:>10(cm), A2: number analyzed (Participants) | 287 | 285 | 282
  After Vac. 1,Swelling:Severe:>10(cm), A2 | 0 | 0 | 0.4
  After Vac. 2, Any Local AEs: number analyzed (Participants) | 264 | 256 | 252
  After Vac. 2, Any Local AEs | 31.1 | 35.9 | 35.7
  After Vac. 2, Pain: Any Severity: number analyzed (Participants) | 263 | 256 | 252
  After Vac. 2, Pain: Any Severity | 27.8 | 30.1 | 31.7
  After Vac. 2, Pain: Mild: number analyzed (Participants) | 263 | 256 | 252
  After Vac. 2, Pain: Mild | 23.6 | 25.8 | 27.8
  After Vac. 2, Pain: Moderate: number analyzed (Participants) | 263 | 256 | 252
  After Vac. 2, Pain: Moderate | 3.4 | 3.5 | 2.8
  After Vac. 2, Pain: Severe: number analyzed (Participants) | 263 | 256 | 252
  After Vac. 2, Pain: Severe | 0.8 | 0.8 | 1.2
  After Vac. 2, Erythema: Any Severity: number analyzed (Participants) | 261 | 256 | 252
  After Vac. 2, Erythema: Any Severity | 12.3 | 14.5 | 13.1
  After Vac. 2,Erythema:Mild:2.5-5(cm): number analyzed (Participants) | 261 | 256 | 252
  After Vac. 2,Erythema:Mild:2.5-5(cm) | 10.7 | 10.5 | 10.7
  After Vac. 2,Erythema:Moderate:>5-<=10(cm): number analyzed (Participants) | 261 | 256 | 252
  After Vac. 2,Erythema:Moderate:>5-<=10(cm) | 1.1 | 3.1 | 2.4
  After Vac. 2,Erythema:Severe:>10(cm): number analyzed (Participants) | 261 | 256 | 252
  After Vac. 2,Erythema:Severe:>10(cm) | 0.4 | 0 | 0
  After Vac. 2, Erythema: Missing Severity: number analyzed (Participants) | 261 | 256 | 252
  After Vac. 2, Erythema: Missing Severity | 0 | 0.8 | 0
  After Vac. 2, Swelling: Any Severity: number analyzed (Participants) | 262 | 256 | 252
  After Vac. 2, Swelling: Any Severity | 2.7 | 5.9 | 5.6
  After Vac. 2,Swelling:Mild:2.5-5(cm): number analyzed (Participants) | 262 | 256 | 252
  After Vac. 2,Swelling:Mild:2.5-5(cm) | 2.3 | 4.3 | 4.8
  After Vac. 2,Swelling:Moderate:>5-<=10(cm): number analyzed (Participants) | 262 | 256 | 252
  After Vac. 2,Swelling:Moderate:>5-<=10(cm) | 0.4 | 1.6 | 0.8
  After Vac. 3, Any Local AEs: number analyzed (Participants) | 237 | 230 | 227
  After Vac. 3, Any Local AEs | 27.8 | 10.4 | 10.6
  After Vac. 3, Pain: Any Severity: number analyzed (Participants) | 237 | 230 | 227
  After Vac. 3, Pain: Any Severity | 24.9 | 10.4 | 9.7
  After Vac. 3, Pain: Mild: number analyzed (Participants) | 237 | 230 | 227
  After Vac. 3, Pain: Mild | 20.3 | 9.1 | 7.9
  After Vac. 3, Pain: Moderate: number analyzed (Participants) | 237 | 230 | 227
  After Vac. 3, Pain: Moderate | 4.2 | 0.9 | 0.9
  After Vac. 3, Pain: Severe: number analyzed (Participants) | 237 | 230 | 227
  After Vac. 3, Pain: Severe | 0.4 | 0.4 | 0.9
  After Vac. 3, Erythema: Any Severity: number analyzed (Participants) | 236 | 229 | 226
  After Vac. 3, Erythema: Any Severity | 9.7 | 0.4 | 0.9
  After Vac. 3,Erythema:Mild:2.5-5(cm): number analyzed (Participants) | 236 | 229 | 226
  After Vac. 3,Erythema:Mild:2.5-5(cm) | 8.5 | 0 | 0.4
  After Vac. 3,Erythema:Moderate:>5-<=10(cm): number analyzed (Participants) | 236 | 229 | 226
  After Vac. 3,Erythema:Moderate:>5-<=10(cm) | 0.4 | 0.4 | 0
  After Vac. 3,Erythema:Severe:>10(cm): number analyzed (Participants) | 236 | 229 | 226
  After Vac. 3,Erythema:Severe:>10(cm) | 0 | 0 | 0.4
  After Vac. 3, Erythema: Missing Severity: number analyzed (Participants) | 236 | 229 | 226
  After Vac. 3, Erythema: Missing Severity | 0.8 | 0 | 0
  After Vac. 3, Swelling: Any Severity: number analyzed (Participants) | 236 | 230 | 227
  After Vac. 3, Swelling: Any Severity | 4.2 | 0 | 0
  After Vac. 3,Swelling:Mild:2.5-5(cm): number analyzed (Participants) | 236 | 230 | 227
  After Vac. 3,Swelling:Mild:2.5-5(cm) | 3.4 | 0 | 0
  After Vac. 3, Swelling: Missing Severity: number analyzed (Participants) | 236 | 230 | 227
  After Vac. 3, Swelling: Missing Severity | 0.8 | 0 | 0

9. Secondary Outcome: Percentage of Participants With Solicited Systemic Adverse Events Following Each Vaccination Dose by Severity
Description: Solicited systemic AEs (fever, headache, asthenia, malaise, and myalgia) recorded from participant's-diary. Severity grades for headache are grade 0 (none), 1 (mild: no interference with daily activity), 2 (moderate: interference with daily activity with or without treatment) and 3 (severe: prevents normal activity with or without treatment). Severity grades for asthenia, malaise and myalgia is grade 0 (none), 1 (mild: no interference with daily activity), 2 (moderate: interference with daily activity), 3 (severe: prevents daily activity). Fever is defined as greater than or equal to 38º C or 100.4º C. Fever was excluded from the overall count as no severity grading was applied for it. Percentages were rounded off for each category.
Time Frame: Within 14 Days of each Vaccination (day of vaccination + 13 days)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: YF-17D + Placebo/TDV/TDV | Group 2: TDV + Placebo/TDV/YF-17D | Group 3: TDV + YF-17D/TDV/Placebo
Number analyzed (Participants) | 300 | 300 | 300
percentage of participants
  After Vaccination 1, Any Systemic AEs: number analyzed (Participants) | 289 | 285 | 282
  After Vaccination 1, Any Systemic AEs | 43.6 | 49.8 | 51.8
  After Vaccination 1, Headache: Any Severity: number analyzed (Participants) | 289 | 285 | 281
  After Vaccination 1, Headache: Any Severity | 31.8 | 33.0 | 39.9
  After Vaccination 1, Headache: Mild: number analyzed (Participants) | 289 | 285 | 281
  After Vaccination 1, Headache: Mild | 21.5 | 22.5 | 26.0
  After Vaccination 1, Headache: Moderate: number analyzed (Participants) | 289 | 285 | 281
  After Vaccination 1, Headache: Moderate | 8.7 | 8.4 | 9.3
  After Vaccination 1, Headache: Severe: number analyzed (Participants) | 289 | 285 | 281
  After Vaccination 1, Headache: Severe | 1.7 | 2.1 | 4.6
  After Vaccination 1, Asthenia: Any Severity: number analyzed (Participants) | 289 | 285 | 281
  After Vaccination 1, Asthenia: Any Severity | 17.6 | 21.1 | 20.3
  After Vaccination 1, Asthenia: Mild: number analyzed (Participants) | 289 | 285 | 281
  After Vaccination 1, Asthenia: Mild | 10.0 | 11.2 | 13.9
  After Vaccination 1, Asthenia: Moderate: number analyzed (Participants) | 289 | 285 | 281
  After Vaccination 1, Asthenia: Moderate | 5.5 | 7.7 | 4.6
  After Vaccination 1, Asthenia: Severe: number analyzed (Participants) | 289 | 285 | 281
  After Vaccination 1, Asthenia: Severe | 2.1 | 2.1 | 1.8
  After Vaccination 1, Malaise: Any Severity: number analyzed (Participants) | 289 | 285 | 282
  After Vaccination 1, Malaise: Any Severity | 20.8 | 20.7 | 24.5
  After Vaccination 1, Malaise: Mild: number analyzed (Participants) | 289 | 285 | 282
  After Vaccination 1, Malaise: Mild | 12.8 | 11.6 | 13.8
  After Vaccination 1, Malaise: Moderate: number analyzed (Participants) | 289 | 285 | 282
  After Vaccination 1, Malaise: Moderate | 6.2 | 4.6 | 8.5
  After Vaccination 1, Malaise: Severe: number analyzed (Participants) | 289 | 285 | 282
  After Vaccination 1, Malaise: Severe | 1.7 | 4.6 | 2.1
  After Vaccination 1, Myalgia: Any Severity: number analyzed (Participants) | 289 | 285 | 282
  After Vaccination 1, Myalgia: Any Severity | 23.2 | 29.5 | 29.4
  After Vaccination 1, Myalgia: Mild: number analyzed (Participants) | 289 | 285 | 282
  After Vaccination 1, Myalgia: Mild | 15.6 | 19.6 | 19.1
  After Vaccination 1, Myalgia: Moderate: number analyzed (Participants) | 289 | 285 | 282
  After Vaccination 1, Myalgia: Moderate | 5.5 | 7.0 | 8.5
  After Vaccination 1, Myalgia: Severe: number analyzed (Participants) | 289 | 285 | 282
  After Vaccination 1, Myalgia: Severe | 2.1 | 2.8 | 1.8
  After Vaccination 1, Fever: Any Severity: number analyzed (Participants) | 288 | 281 | 279
  After Vaccination 1, Fever: Any Severity | 1.4 | 6.0 | 1.1
  After Vaccination 1,Fever:38.0-<38.5: number analyzed (Participants) | 288 | 281 | 279
  After Vaccination 1,Fever:38.0-<38.5 | 0.3 | 3.6 | 0.4
  After Vaccination 1,Fever:38.5-<39.0: number analyzed (Participants) | 288 | 281 | 279
  After Vaccination 1,Fever:38.5-<39.0 | 0.3 | 1.8 | 0.7
  After Vaccination 1,Fever:39.0-<39.5: number analyzed (Participants) | 288 | 281 | 279
  After Vaccination 1,Fever:39.0-<39.5 | 0.3 | 0.4 | 0
  After Vaccination 1,Fever:39.5-<40.0: number analyzed (Participants) | 288 | 281 | 279
  After Vaccination 1,Fever:39.5-<40.0 | 0 | 0.4 | 0
  After Vaccination 1,Fever:≥41.0: number analyzed (Participants) | 288 | 281 | 279
  After Vaccination 1,Fever:≥41.0 | 0.3 | 0 | 0
  After Vaccination 2, Any Systemic AEs: number analyzed (Participants) | 264 | 256 | 252
  After Vaccination 2, Any Systemic AEs | 33.3 | 29.3 | 31.7
  After Vaccination 2, Headache: Any Severity: number analyzed (Participants) | 264 | 256 | 252
  After Vaccination 2, Headache: Any Severity | 22.7 | 15.6 | 21.0
  After Vaccination 2, Headache: Mild: number analyzed (Participants) | 264 | 256 | 252
  After Vaccination 2, Headache: Mild | 13.3 | 10.2 | 11.9
  After Vaccination 2, Headache: Moderate: number analyzed (Participants) | 264 | 256 | 252
  After Vaccination 2, Headache: Moderate | 6.4 | 4.3 | 7.1
  After Vaccination 2, Headache: Severe: number analyzed (Participants) | 264 | 256 | 252
  After Vaccination 2, Headache: Severe | 3.0 | 1.2 | 2.0
  After Vaccination 2, Asthenia: Any Severity: number analyzed (Participants) | 264 | 256 | 252
  After Vaccination 2, Asthenia: Any Severity | 13.3 | 8.6 | 11.5
  After Vaccination 2, Asthenia: Mild: number analyzed (Participants) | 264 | 256 | 252
  After Vaccination 2, Asthenia: Mild | 8.3 | 2.7 | 6.7
  After Vaccination 2, Asthenia: Moderate: number analyzed (Participants) | 264 | 256 | 252
  After Vaccination 2, Asthenia: Moderate | 3.8 | 4.3 | 2.4
  After Vaccination 2, Asthenia: Severe: number analyzed (Participants) | 264 | 256 | 252
  After Vaccination 2, Asthenia: Severe | 1.1 | 1.6 | 2.4
  After Vaccination 2, Malaise: Any Severity: number analyzed (Participants) | 264 | 256 | 252
  After Vaccination 2, Malaise: Any Severity | 14.0 | 9.8 | 9.9
  After Vaccination 2, Malaise: Mild: number analyzed (Participants) | 264 | 256 | 252
  After Vaccination 2, Malaise: Mild | 7.6 | 4.3 | 4.4
  After Vaccination 2, Malaise: Moderate: number analyzed (Participants) | 264 | 256 | 252
  After Vaccination 2, Malaise: Moderate | 4.5 | 4.3 | 4.0
  After Vaccination 2, Malaise: Severe: number analyzed (Participants) | 264 | 256 | 252
  After Vaccination 2, Malaise: Severe | 1.9 | 1.2 | 1.6
  After Vaccination 2, Myalgia: Any Severity: number analyzed (Participants) | 264 | 256 | 252
  After Vaccination 2, Myalgia: Any Severity | 20.8 | 18.8 | 20.2
  After Vaccination 2, Myalgia: Mild: number analyzed (Participants) | 264 | 256 | 252
  After Vaccination 2, Myalgia: Mild | 14.4 | 13.3 | 12.3
  After Vaccination 2, Myalgia: Moderate: number analyzed (Participants) | 264 | 256 | 252
  After Vaccination 2, Myalgia: Moderate | 5.3 | 4.3 | 5.2
  After Vaccination 2, Myalgia: Severe: number analyzed (Participants) | 264 | 256 | 252
  After Vaccination 2, Myalgia: Severe | 1.1 | 1.2 | 2.8
  After Vaccination 2, Fever: Any Severity: number analyzed (Participants) | 260 | 250 | 248
  After Vaccination 2, Fever: Any Severity | 3.1 | 1.2 | 1.2
  After Vaccination 2,Fever:38.0-<38.5: number analyzed (Participants) | 260 | 250 | 248
  After Vaccination 2,Fever:38.0-<38.5 | 1.5 | 0.4 | 0.4
  After Vaccination 2,Fever:38.5-<39.0: number analyzed (Participants) | 260 | 250 | 248
  After Vaccination 2,Fever:38.5-<39.0 | 1.2 | 0.8 | 0.4
  After Vaccination 2,Fever:39.0-<39.5: number analyzed (Participants) | 260 | 250 | 248
  After Vaccination 2,Fever:39.0-<39.5 | 0.4 | 0 | 0
  After Vaccination 2,Fever:39.5-<40.0: number analyzed (Participants) | 260 | 250 | 248
  After Vaccination 2,Fever:39.5-<40.0 | 0 | 0 | 0.4
  After Vaccination 3, Any Systemic AEs: number analyzed (Participants) | 238 | 230 | 228
  After Vaccination 3, Any Systemic AEs | 24.4 | 27.4 | 22.8
  After Vaccination 3, Headache: Any Severity: number analyzed (Participants) | 238 | 230 | 228
  After Vaccination 3, Headache: Any Severity | 17.2 | 17.4 | 20.2
  After Vaccination 3, Headache: Mild: number analyzed (Participants) | 238 | 230 | 228
  After Vaccination 3, Headache: Mild | 10.1 | 11.3 | 13.6
  After Vaccination 3, Headache: Moderate: number analyzed (Participants) | 238 | 230 | 228
  After Vaccination 3, Headache: Moderate | 6.3 | 4.8 | 4.8
  After Vaccination 3, Headache: Severe: number analyzed (Participants) | 238 | 230 | 228
  After Vaccination 3, Headache: Severe | 0.8 | 1.3 | 1.8
  After Vaccination 3, Asthenia: Any Severity: number analyzed (Participants) | 238 | 230 | 228
  After Vaccination 3, Asthenia: Any Severity | 10.5 | 9.1 | 7.0
  After Vaccination 3, Asthenia: Mild: number analyzed (Participants) | 238 | 230 | 228
  After Vaccination 3, Asthenia: Mild | 6.3 | 7.4 | 3.9
  After Vaccination 3, Asthenia: Moderate: number analyzed (Participants) | 238 | 230 | 228
  After Vaccination 3, Asthenia: Moderate | 3.8 | 1.7 | 2.6
  After Vaccination 3, Asthenia: Severe: number analyzed (Participants) | 238 | 230 | 228
  After Vaccination 3, Asthenia: Severe | 0.4 | 0 | 0.4
  After Vaccination 3, Malaise: Any Severity: number analyzed (Participants) | 238 | 230 | 228
  After Vaccination 3, Malaise: Any Severity | 11.3 | 13.5 | 11.4
  After Vaccination 3, Malaise: Mild: number analyzed (Participants) | 238 | 230 | 228
  After Vaccination 3, Malaise: Mild | 6.3 | 9.1 | 7.9
  After Vaccination 3, Malaise: Moderate: number analyzed (Participants) | 238 | 230 | 228
  After Vaccination 3, Malaise: Moderate | 3.8 | 3.5 | 2.6
  After Vaccination 3, Malaise: Severe: number analyzed (Participants) | 238 | 230 | 228
  After Vaccination 3, Malaise: Severe | 1.3 | 0.9 | 0.9
  After Vaccination 3, Myalgia: Any Severity: number analyzed (Participants) | 238 | 230 | 228
  After Vaccination 3, Myalgia: Any Severity | 12.6 | 12.2 | 7.9
  After Vaccination 3, Myalgia: Mild: number analyzed (Participants) | 238 | 230 | 228
  After Vaccination 3, Myalgia: Mild | 7.6 | 7.8 | 4.8
  After Vaccination 3, Myalgia: Moderate: number analyzed (Participants) | 238 | 230 | 228
  After Vaccination 3, Myalgia: Moderate | 3.8 | 3.9 | 2.6
  After Vaccination 3, Myalgia: Severe: number analyzed (Participants) | 238 | 230 | 228
  After Vaccination 3, Myalgia: Severe | 1.3 | 0.4 | 0.4
  After Vaccination 3, Fever: Any Severity: number analyzed (Participants) | 234 | 228 | 227
  After Vaccination 3, Fever: Any Severity | 1.3 | 0 | 1.3
  After Vaccination 3,Fever:38.0-<38.5: number analyzed (Participants) | 234 | 228 | 227
  After Vaccination 3,Fever:38.0-<38.5 | 0.9 | 0 | 0.9
  After Vaccination 3,Fever:38.5-<39.0: number analyzed (Participants) | 234 | 228 | 227
  After Vaccination 3,Fever:38.5-<39.0 | 0.4 | 0 | 0
  After Vaccination 3,Fever:39.0-<39.5: number analyzed (Participants) | 234 | 228 | 227
  After Vaccination 3,Fever:39.0-<39.5 | 0 | 0 | 0.4

10. Secondary Outcome: Percentage of Participants With Any Unsolicited Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a trial vaccine; it does not necessarily have to have a causal relationship with trial vaccine administration.
Time Frame: Within 28 days (day of vaccination + 27 days) after each vaccination
Population: Safety Set included all randomized participants who received at least 1 dose of the trial vaccines. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: YF-17D + Placebo/TDV/TDV | Group 2: TDV + Placebo/TDV/YF-17D | Group 3: TDV + YF-17D/TDV/Placebo
Number analyzed (Participants) | 300 | 300 | 300
percentage of participants
  After First Vaccination | 11.7 | 17.3 | 14.0
  After Second Vaccination: number analyzed (Participants) | 273 | 270 | 264
  After Second Vaccination | 8.8 | 10.4 | 9.1
  After Third Vaccination: number analyzed (Participants) | 248 | 241 | 233
  After Third Vaccination | 4.4 | 5.4 | 4.7

11. Secondary Outcome: Percentage of Participants With Medically Attended Adverse Events (MAAEs)
Description: MAAEs are defined as AEs leading to an unscheduled visit to or by a healthcare professional including visits to an emergency department, but not fulfilling seriousness criteria.
Time Frame: From first vaccination (Day 1) through end of study (Day 360)
Population: Safety Set included all randomized participants who received at least 1 dose of the trial vaccines.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: YF-17D + Placebo/TDV/TDV | Group 2: TDV + Placebo/TDV/YF-17D | Group 3: TDV + YF-17D/TDV/Placebo
Number analyzed (Participants) | 300 | 300 | 300
percentage of participants | 14.3 | 15.3 | 15.3

12. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, leads to a congenital anomaly/birth defect in the offspring of a participant, is an important medical event that may require intervention to prevent any of the above mentioned criteria and/or may expose the subject to danger, even though the event is not immediately life threatening or fatal or does not result in hospitalization.
Time Frame: From first vaccination (Day 1) through end of study (Day 360)
Population: Safety Set included all randomized participants who received at least 1 dose of the trial vaccines.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: YF-17D + Placebo/TDV/TDV | Group 2: TDV + Placebo/TDV/YF-17D | Group 3: TDV + YF-17D/TDV/Placebo
Number analyzed (Participants) | 300 | 300 | 300
percentage of participants | 4.3 | 3.3 | 2.3

ADVERSE EVENTS:
Time Frame: All-Cause Mortality and Serious Adverse Events: From first vaccination (Day 1) through end of study (Day 360); Other Adverse Events: From any vaccination (Day 1, Day 90, and Day 180) up to 28 days post vaccination.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Group 1: YF-17D + Placebo/TDV/TDV | Group 2: TDV + Placebo/TDV/YF-17D | Group 3: TDV + YF-17D/TDV/Placebo
All-Cause Mortality (participants affected / at risk) | 0/300 | 1/300 | 1/300
Serious Adverse Events (participants affected / at risk) | 13/300 | 10/300 | 7/300
Other Adverse Events (participants affected / at risk) | 11/300 | 23/300 | 19/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: YF-17D + Placebo/TDV/TDV (N=300) | Group 2: TDV + Placebo/TDV/YF-17D (N=300) | Group 3: TDV + YF-17D/TDV/Placebo (N=300)
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Megacolon (Gastrointestinal disorders) | 0 | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Allergy to arthropod sting (Immune system disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 2
Abscess intestinal (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Aesthesioneuroblast oma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 1
Drug abuse (Psychiatric disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Organ donor (Social circumstances) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: YF-17D + Placebo/TDV/TDV (N=300) | Group 2: TDV + Placebo/TDV/YF-17D (N=300) | Group 3: TDV + YF-17D/TDV/Placebo (N=300)
Injection site bruising (General disorders) | 4 | 5 | 10
Injection site pruritus (General disorders) | 3 | 7 | 8
Upper respiratory tract infection (Infections and infestations) | 6 | 13 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT03342898/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT03342898/SAP_001.pdf